CLINICAL TRIAL: NCT04622098
Title: Prevalence of Sub-epithelial Lesions Among Patients Undergoing EGDs in Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Collaborators: Mansoura University Hospital (Other); Menoufia University (Other); Al-Azhar University (Other); Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Salah Zaghloul, Doctor, Kafrelsheikh University
Other Study IDs: 135/2020
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2020-11

CONDITIONS: Esophageal Neoplasms; Gastric Neoplasm; Duodenal Neoplasms
Keywords: sub-epithelial lesions; esophagogastrodudenoscopy; EUS FNA/FNB
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Duodenal Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample for routine laboratory inverstigations tissue sample from the SEL if indicated or gross excisional sample post surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with SEL: Any patient with detected sub-epithelial lesion during upper endoscopy either symptomatized or accidently discovered.
  Patients diagnosed by EUS, CT scan or surgically removed lesions.
  Interventions: Procedure: Endoscopic ultrasound

INTERVENTIONS:
Procedure: Endoscopic ultrasound — this is an endoscopic procedure for the assessment of the lesions, the following will be recorded:
  1. the tumor location,
  2. layer of origin,
  3. maximal diameter,
  4. regularity of extraluminal border,
  5. echopattern,
  6. presence of cystic spaces or echogenic foci.
  Other Names: CT

SUMMARY:
Subepithelial lesions (SEL) are incidentally observed in the stomach of about 0.3% of middle-aged men and women; half of these are neoplastic. The incidence of subepithelial tumors (SET) of gastrointestinal (GI) origin has risen twofold to fivefold within the past 30 years.The etiology of most SMTs cannot easily be determined by endoscopy. So, we aim to estimate the prevalence and types of sub-epithelial lesions among patients undergoing EGDs in Egypt.

DETAILED DESCRIPTION:
Worldwide, the gastrointestinal (GI) tract is the organ system with the highest cancer incidence (20.5% of all new cases) and annual mortality (22% = 1.81 Mio). Early endoscopic detection and resection has led to improved survival rates for colorectal and gastric cancer, especially for gastric cancer in Japan, where more than 70% are now detected as early gastric cancer. Subepithelial lesions (SELs) of the GI tract are tumors that originate from the muscularis mucosa, submucosa, or muscularis propria. The term subepithelial lesion is preferred to the term submucosal tumor, which should be reserved for those that originate from the submucosal layer. SELs are most commonly found in the stomach, as often as 1 in every 300 endoscopies. The majority of these tumors are benign, with fewer than 15% found to be malignant at presentation.

Subepithelial lesions (SEL) are incidentally observed in the stomach of about 0.3% of middle-aged men and women; half of these are neoplastic. The incidence of subepithelial tumors (SET) of gastrointestinal (GI) origin has risen twofold to fivefold within the past 30 years.

According to the Korea EUS Study Group (unpublished data), the prevalence of gastric SETs, detected routine esophagogastroduodenoscopy, in Korea is 3.1%.

The etiology of most SMTs cannot easily be determined by endoscopy. Subepithelial lesions are those located beneath the epithelium and originate from any layer of the gastrointestinal wall. EUS is the best imaging modality to assess gastrointestinal subepithelial lesions and can be used for EUS guided tissue sampling, in addition to diagnostic imaging of the nodule. It helps to distinguish extrinsic lesions from intramural ones based on the originating layer, echogenicity and tissue acquisition to reach an accurate diagnosis. In clinical practice, cytological and immunocytochemical results determine the final diagnosis. EUS is superior to other imaging modalities (CT, magnetic resonance imaging) in characterizing small (<2 cm) lesions.

NCCN guideline on GISTs recommends resection of all symptomatic lesions, any lesions that are ≥2 cm, or lesions that have high risk features under EUS. Annual surveillance is recommended for low risk GISTs. Neuroendocrine tumours (NET) , meanwhile, has higher malignant potentials. Some investigators advocate resecting all visible lesions. The minimal approach should be to resect tumors ≥1 cm in diameter. NET require surveillance similar if not more stringent than GIST.

Endoscopic mucosal forceps biopsy is the standard procedures for establishing diagnoses in patients with GI tumors. However, the false negative rate of endoscopic mucosal forceps biopsy can be as high as 50%. Possible reasons for this false negative rate include infiltrative and stenotic diseases as well as lesions in submucosal locations, such as lymphoma.

Because of their subepithelial location, biopsies with endoscopic forceps often fail to provide diagnostic tissues. Thus, further imaging and sampling techniques (often with EUS) often are used to characterize these lesions especially in large lesions.

Study objectives:

1. Primary Objectives:

   Estimating the prevalence and types of sub-epithelial lesions among patients undergoing EGDs in Egypt.
2. Secondary objectives:

Determining the real predominance of sub-epithelial lesions considering sex and age differences.

Investigating the geographic distribution in relation to the diagnosis of the lesions.

Detecting the commonest sites for the sub-epithelial lesions. Recording the symptomology related to each type.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with detected sub-epithelial lesion during upper endoscopy either symptomatized or accidently discovered.
2. Patients diagnosed by EUS, CT scan or surgically removed lesions.

Exclusion Criteria:

1. Patients missing follow up to reach a sure diagnosis for the lesions.
2. Patients unfit for endoscopic procedures.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presented to endoscopy units participating in the study and in need for upper endoscopy will be given informed written consent to participate in the study. Possible complications will be described clearly to the patients before the endoscopic procedure. Complete medical history will be recorded specially symptoms suggesting GIT bleeding as hematemesis, melena, or manifestations of anemia. Symptoms suggesting malignancy as weight loss, anorexia, history of previous malignancies will be recorded. Past history of endoscopic procedures, of having previous GIT troubles and of any chronic medical illness or medications will be recorded. Vital signs will be taken for the patients before beginning the endoscopic procedure and after being evaluated by an anesthetist.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Estimating the prevalence and types of sub-epithelial lesions among patients undergoing EGDs in Egypt. | 6 months
  prevalence rate

SECONDARY OUTCOMES:
characterization of SEL in Egypt | one year
  correlation to demographic data

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hwang JH, Rulyak SD, Kimmey MB; American Gastroenterological Association Institute. American Gastroenterological Association Institute technical review on the management of gastric subepithelial masses. Gastroenterology. 2006 Jun;130(7):2217-28. doi: 10.1053/j.gastro.2006.04.033. PMID 16762644
- [Result] Standards of Practice Committee; Faulx AL, Kothari S, Acosta RD, Agrawal D, Bruining DH, Chandrasekhara V, Eloubeidi MA, Fanelli RD, Gurudu SR, Khashab MA, Lightdale JR, Muthusamy VR, Shaukat A, Qumseya BJ, Wang A, Wani SB, Yang J, DeWitt JM. The role of endoscopy in subepithelial lesions of the GI tract. Gastrointest Endosc. 2017 Jun;85(6):1117-1132. doi: 10.1016/j.gie.2017.02.022. Epub 2017 Apr 3. No abstract available. PMID 28385194
- [Result] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Result] Papanikolaou IS, Triantafyllou K, Kourikou A, Rosch T. Endoscopic ultrasonography for gastric submucosal lesions. World J Gastrointest Endosc. 2011 May 16;3(5):86-94. doi: 10.4253/wjge.v3.i5.86. PMID 21772939
- [Result] Polkowski M. Endoscopic ultrasound and endoscopic ultrasound-guided fine-needle biopsy for the diagnosis of malignant submucosal tumors. Endoscopy. 2005 Jul;37(7):635-45. doi: 10.1055/s-2005-861422. No abstract available. PMID 16010608
- [Result] Hedenbro JL, Ekelund M, Wetterberg P. Endoscopic diagnosis of submucosal gastric lesions. The results after routine endoscopy. Surg Endosc. 1991;5(1):20-3. doi: 10.1007/BF00591381. PMID 1871670
- [Result] Nishida T, Kawai N, Yamaguchi S, Nishida Y. Submucosal tumors: comprehensive guide for the diagnosis and therapy of gastrointestinal submucosal tumors. Dig Endosc. 2013 Sep;25(5):479-89. doi: 10.1111/den.12149. Epub 2013 Jul 31. PMID 23902569
- [Result] Wiech T, Walch A, Werner M. Histopathological classification of nonneoplastic and neoplastic gastrointestinal submucosal lesions. Endoscopy. 2005 Jul;37(7):630-4. doi: 10.1055/s-2005-870127. PMID 16010607
- [Result] Park EY, Kim GH. Diagnosis of Gastric Subepithelial Tumors Using Endoscopic Ultrasonography or Abdominopelvic Computed Tomography: Which is Better? Clin Endosc. 2019 Nov;52(6):519-520. doi: 10.5946/ce.2019.188. Epub 2019 Nov 14. No abstract available. PMID 31722518
- [Result] Mathew, Madhu MD1; Mbachi, Chimezie MD1; Desai, Parth M. DO1; Salazar, Miguel MD2; Vohra, Ishaan MD1; Wang, Yuchen MD2; Gandhi, Seema MD3; Attar, Bashar M. MD, PhD1 2893 Epidemiology of Sub-Epithelial Gastrointestinal Lesions and Factors Influencing Their Tissue Yield by EUS Guided Sampling in a Predominantly African-American and Hispanic Population at a Tertiary Care County Hospital, The American Journal of Gastroenterology: October 2019 - Volume 114 - Issue - p S1584 doi: 10.14309/01.ajg.0000601104.52032.6f
- [Result] Okten RS, Kacar S, Kucukay F, Sasmaz N, Cumhur T. Gastric subepithelial masses: evaluation of multidetector CT (multiplanar reconstruction and virtual gastroscopy) versus endoscopic ultrasonography. Abdom Imaging. 2012 Aug;37(4):519-30. doi: 10.1007/s00261-011-9791-0. PMID 21822967
- [Result] Demetri GD, von Mehren M, Antonescu CR, DeMatteo RP, Ganjoo KN, Maki RG, Pisters PW, Raut CP, Riedel RF, Schuetze S, Sundar HM, Trent JC, Wayne JD. NCCN Task Force report: update on the management of patients with gastrointestinal stromal tumors. J Natl Compr Canc Netw. 2010 Apr;8 Suppl 2(0 2):S1-41; quiz S42-4. doi: 10.6004/jnccn.2010.0116. PMID 20457867
- [Result] Delle Fave G, O'Toole D, Sundin A, Taal B, Ferolla P, Ramage JK, Ferone D, Ito T, Weber W, Zheng-Pei Z, De Herder WW, Pascher A, Ruszniewski P; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for Gastroduodenal Neuroendocrine Neoplasms. Neuroendocrinology. 2016;103(2):119-24. doi: 10.1159/000443168. Epub 2016 Jan 19. No abstract available. PMID 26784901
- [Result] Ramage JK, De Herder WW, Delle Fave G, Ferolla P, Ferone D, Ito T, Ruszniewski P, Sundin A, Weber W, Zheng-Pei Z, Taal B, Pascher A; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for Colorectal Neuroendocrine Neoplasms. Neuroendocrinology. 2016;103(2):139-43. doi: 10.1159/000443166. Epub 2016 Jan 5. No abstract available. PMID 26730835
- [Result] Palazzo L, Landi B, Cellier C, Cuillerier E, Roseau G, Barbier JP. Endosonographic features predictive of benign and malignant gastrointestinal stromal cell tumours. Gut. 2000 Jan;46(1):88-92. doi: 10.1136/gut.46.1.88. PMID 10601061
- [Result] ASGE Standards of Practice Committee; Chandrasekhara V, Khashab MA, Muthusamy VR, Acosta RD, Agrawal D, Bruining DH, Eloubeidi MA, Fanelli RD, Faulx AL, Gurudu SR, Kothari S, Lightdale JR, Qumseya BJ, Shaukat A, Wang A, Wani SB, Yang J, DeWitt JM. Adverse events associated with ERCP. Gastrointest Endosc. 2017 Jan;85(1):32-47. doi: 10.1016/j.gie.2016.06.051. Epub 2016 Aug 18. No abstract available. PMID 27546389